CLINICAL TRIAL: NCT04292210
Title: Evaluating Patient Safety And Ease Of Use Of A Novel Connection-Assist Device For Peritoneal Dialysis
Brief Title: Human Factors Validation Testing for the Peripal System; a Manual Connection Assist Device for Peritoneal Dialysis Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peripal AG (Industry)
Collaborators: Swiss Federal Institute of Technology (Other); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS ID :235715
Record Dates: First submitted 2020-02-19; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: End Stage Renal Failure on Dialysis; End Stage Renal Disease on Dialysis; Renal Failure; Peritoneal Dialysis; Renal Replacement Therapy
Keywords: patient safety; usability study; connection-assist device; ease of use; peritoneal dialysis; NASA Task Load Index; renal replacement therapy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: The growth in the RRT population is primary in the elderly age group, a population with a high frailty and comorbidity burden. Facilitating PD in this group of patients requires improved PD technology with greater accessibility tailored to patient needs. It is proposed that by making PD treatment simpler, more standardized and better protected from infections, patient access to PD could be increased significantly. Following evaluation of specific barriers to the use of PD including feedback from established PD patients, a novel connection-assist device has been developed.
  As part of the CE marking authorization, the connection device has been evaluated for safety and ease of use in a study at University Hospitals Birmingham NHS Foundation Trust involving 24 patients and carers.
Masking Description: The training consisted of two cycles in which the moderator guided the subject and three cycles in which the subject guided the moderator through the complete handling of the device.
  For each subject, one moderator and one observer were involved in the study. The moderator was the interface between the subject and the device both in training and in testing. This person was employed by an external agency to avoid any influence on the subject.
  The observer saw the handling with the help of a live feed from a separate room. He evaluated the handling steps in the categories of "safe use" and "use error" according to IEC 62366-1 (2015). For each use error, the observer described the observed situation from his point of view.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPD handling (Experimental): A connecting device simplifying the steps during a cycle of Peritoneal dialysis. Instead of directly doing a manual connection and manually breaking a frangible, the device assist in connecting and breaking the frangible.
  This study was done demonstrating a continuous ambulatory peritoneal dialysis (CAPD)
  Interventions: Device: Perisafe

INTERVENTIONS:
Device: Perisafe — A medical device simplifying the connection of tubing as well as breaking of the frangible which is done in a sterile environment with the help of levers and buttons.

SUMMARY:
It is estimated that there are currently over 3 million patients receiving dialysis treatment worldwide. With effective pre-dialysis counselling, a majority of patients choose the home-based therapy peritoneal dialysis (PD) but only approximately 11% of prevalent dialysis patients use this modality. Connection-assist devices can overcome the challenges posed by decreased manual dexterity and/or visual acuity, and can allow more patients to be treated with home-based therapies. As part of the CE marking authorization, a connection device has been evaluated for safety and ease of use in a usability study.

DETAILED DESCRIPTION:
The growth in the renal replacement therapy population is primaryly in the elderly age group, a population with a high frailty and comorbidity burden. Facilitating PD in this group of patients requires improved PD technology with greater accessibility tailored to patient needs. Following evaluation of specific barriers to the use of PD including feedback from established PD patients, a novel connection-assist device has been developed.

As part of the CE marking authorization, the connection device has been evaluated for safety and ease of use in a study at University Hospitals Birmingham NHS Foundation Trust involving 24 patients and carers.

The evaluated device is designed to assist peritoneal dialysis patients performing their daily dialysis treatment either for APD or for CAPD. The device facilitates the connection and disconnection of the dialysis line to the PD catheter transfer set. The connections are performed inside the device in a protected area, and the patient does not need to touch the transfer set or the dialysis line while they are unprotected. In addition, the breaking of the dialysis line frangible and the clamping of the dialysis line are replaced by pushing a button.

The operating procedure of the device consists of multiple tasks including preparing and loading the transfer set and dialysis line into the device, performing the handling steps related to the PD therapy with the device and finally unloading the used material from the device. Each task comprises several handling steps. During the study, the operating procedure with the device was simulated and the subjects were connected to a dummy catheter, which was attached to an apron.

This study recruited established PD patients and carers involved in the delivery of PD. Carers included healthcare professionals and lay carers.

The study design was divided into three one hour long parts. Firstly, a training session introduced the operation of the device. Secondly, a break of one hour allowed relaxation and recovery. Thirdly, a test was carried out to determine whether the subject could use the device independently with the aid of a quick start guide and the device manual.

The training consisted of two cycles in which the moderator guided the subject and three cycles in which the subject guided the moderator through the complete handling of the device. After the break, the subjects were asked to carry out a complete handling cycle themselves. Subjects could use the quick start guide and the device manual as help. After the unsupported handling cycle, subjects were asked to complete the NASA Task Load Index (N-TLX) questionnaire. In the meantime, the moderator left the room to obtain information on observed use errors. In a final semi-structured interview, the subjects were asked about the reasons for the observed use errors.

For each subject, one moderator and one observer were involved in the study. The moderator was the interface between the subject and the device both in training and in testing. This person was employed by an external agency to avoid any influence on the subject. The observer saw the handling with the help of a live feed from a separate room. He evaluated the handling steps in the categories of "safe use" and "use error" according to IEC 62366-1. For each use error, the observer described the observed situation from his point of view. In addition to evaluating the effectiveness of the task performance, the subjects were interviewed in a semi structured way. Here the observations of technique errors were discussed with the subjects in order to identify the specific causes. In this interview, the subjects were also asked for their feedback on the general ease of use of the device.

In addition, the subjects were asked about the task load in six different dimensions in the standardized N-TLX. Task load is a hypothetical construct that represents the cost incurred by a human operator to achieve a particular level of performance. The dimensions of the N-TLX are mental, physical and temporal demands as well as performance, effort and frustration in the task. Each dimension is evaluated on a 20-point scale. This scale is then transferred to the task load index, which is a scale between 0 and 100 points. To classify the results of the N-TLX, Eitrheim and Fernandes (2016) state "Workload levels below 50 were perceived as acceptable."

ELIGIBILITY:
Fifteen patients and nine carers volunteered in this study, ranging from 23 to 86 years in age and from 0.3 to 24 years in experience in the PD therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and ease of use of a connection device during a continuous ambulatory peritoneal dialysis | 3 hours
  Firstly, a training session introduced the operation of the device. The normal steps of a manual connection and breaking of the frangible is replaced by the levers and the buttons in the device. The connections are thereby done in a 'safe' environment which reduces infection risk. A whole cycle of continuous ambulatory peritoneal dialysis is simulated during each training. Secondly, a break of one hour allowed relaxation and recovery. Thirdly, a test was carried out to determine whether the subject could use the device independently with the aid of a quick start guide and the device manual.
  The training consisted of two cycles in which the moderator guided the subject and three cycles in which the subject guided the moderator through the complete handling of the device.
  Each of the 24 subjects performed 52 handling steps resulting in a total of 1248 evaluated handling steps.
Nasa Task Load Index (N-TLX) | 3 hours
  The operating procedure of the device consists of multiple tasks comprising several handling steps. the subjects were asked about the task load in six different dimensions in the standardized N-TLX. Task load is a hypothetical construct that represents the cost incurred by a human operator to achieve a particular level of performance. The dimensions of the N-TLX are mental, physical and temporal demands as well as performance, effort and frustration in the task. Each dimension is evaluated on a 20-point scale. This scale is then transferred to the task load index, which is a scale between 0 and 100 points. Workload levels below 50 were perceived as acceptable.
Observation of technique | 3 hours.
  Here the observations of technique errors were discussed with the subjects in order to identify the specific causes. In this interview, the subjects were also asked for their feedback on the general ease of use of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Foggensteiner, MD, PhD, Study Chair — National Health Service, United Kingdom; Mirko Meboldt, PhD, Study Chair — ETH; Martin Dubach, Study Chair — Peripal AG; Stephan Hess, Principal Investigator — ETH
Locations (1):
- NIHR Trauma Management MedTech Co-operative, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Evaluating Patient Safety and Ease of use of a Novel Connection-Assist Device for Peritoneal Dialysis — https://www.dovepress.com/evaluating-patient-safety-and-ease-of-use-of-a-novel-connection-assist-peer-reviewed-article-PPA